CLINICAL TRIAL: NCT06393946
Title: Observational Study in Adults With Severe Chronic Rhinosinusitis With Nasal Polyposis (CRSwNP) Treated With Dupilumab in France
Brief Title: Study in Adults With Severe Chronic Rhinosinusitis With Nasal Polyposis Treated With Dupilumab in France
Acronym: OPALE
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17269; U1111-1264-3068 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-04-10; First posted 2024-05-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyposis
Keywords: Real World Evidence (RWE); ENT disease; CRSwNP; Nasal Polyp Syndrome; Dupixent; Surgery
MeSH Terms: conditions — Otorhinolaryngologic Diseases | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dupilumab: The information will be collected during consultation as part of the patient's usual follow-up.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — This study will not administer any treatment, only observe the treatment as prescribed in real world-clinical practice.

SUMMARY:
This is a multicentre, non-interventional, single arm study that aims to describe the treatment patterns in France: patients' characteristics, disease characteristics, prior treatments for Severe chronic rhinosinusitis with nasal polyposis and treatment prescription modalities. As well as to assess the clinical outcome after initiation of dupilumab (Dupixent®) and safety of the product during the two years of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient aged >= 18 years old at the time of the initiation of the treatment with dupilumab (Dupixent®).
* Decision to initiate Dupixent® prior to inclusion in the study, initiation of Dupixent® for severe Chronic rhinosinusitis with nasal polyposis (CRSwNP) maximum 3 months before inclusion.
* Informed consent and willingness to participate.

Exclusion Criteria:

* Conditions or legal situations resulting in impossibility to consent or impacting the interpretation of the results.
* Patient participating in an interventional clinical trial with experimental product at inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with asthma initiating Dupilumab for their Severe chronic rhinosinusitis with nasal polyposis (CRSwNP) according to the prescribing information in France.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics: Age | At baseline (Day 1)
Patient characteristics: Sex | At baseline (Day 1)
Patient characteristics: Weight | At baseline (Day 1)
Patient characteristics: Height | At baseline (Day 1)
Patient characteristics: Type 2 comorbidities | At baseline (Day 1)
  The following patient characteristics will be described: Documented comorbidities associated with type 2 inflammation (asthma + severity, atopic dermatitis, Aspirin Exacerbated Disease (AERD), chronic allergic rhinitis)
Patient characteristics: Medical history | At baseline (Day 1)
  Including CRSwNP history and CRSwNP family history.
Patient characteristics: Lifestyle habits | At baseline (Day 1)
  Including smoking habits
Disease characteristics: CRSwNP duration | At baseline (Day 1)
Disease characteristics: Age at diagnosis of CRSwNP | At baseline (Day 1)
Disease characteristics: Blood Eosinophils | At baseline (Day 1)
  The results of the last test carried out before Dupixent® initiation will be used as baseline, as per standard of care, if available.
Disease characteristics: Total serum IgE | At baseline (Day 1)
  The results of the last test carried out before Dupixent® initiation will be used as baseline, as per standard of care, if available.
Disease characteristics: Anatomopathology | At baseline (Day 1)
  The results of the last exam carried out before Dupixent® initiation will be used as baseline, as per standard of care, if available.
Disease characteristics: Nasal polyps score (NPS) at baseline | At baseline (Day 1)
  The nasal polyps endoscopic score (NPS) assesses length and distribution of polyps, with a score from 0 to 4 for each nostril, maximum bilateral score of 8 points. Meaning lower (0=no polyp) and higher (4=large polyps).
Disease characteristics: Nasal congestion score (NCS) at baseline | At baseline (Day 1)
  The Nasal congestion score (NCS) was assessed on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicating more severity.
Disease characteristics: Rhinorrhea score (anterior/posterior) at baseline | At baseline (Day 1)
  The rhinorrhea scores are scored from 0 ('No symptoms') to 3 ('Severe symptoms'). Where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicating more severity.
Disease characteristics: VAS for CRSwNP symptoms at baseline | At baseline (Day 1)
  The Visual Analog Scale for CRSwNP assesses symptoms, ranging from 0 to 10:
  * mild if VAS between 0 and 3
  * moderate if VAS between > 3 and 7
  * severe if VAS between > 7 and 10.
Disease characteristics: smell test score Visual Analog Scale (VAS) at baseline | At baseline (Day 1)
  Participants value their olfactory function by using the Visual Analogue Scale (VAS), the range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome), where higher score indicated worse thinkable troublesome.
Concomitant and prior medications for CRSwNP or other disease: Number of patients with at least one prior or concomitant SCS | From baseline up to 24 months.
  Number of patients with at least one prior or concomitant Systemic Corticosteroids (SCS)
Concomitant and prior medications for CRSwNP or other disease:Type of prior Systemic Corticosteroids (SCS) per patient | From baseline up to 24 months.
  Prior (resp. concomitant) SCS taken (Prednisone/Prednisolone/Betamethasone/Methylprednisolone)
Concomitant and prior medications for CRSwNP or other disease: Cumulative dose of SCS | From baseline up to 24 months.
  Cumulative dose over the past year
Concomitant and prior medications for CRSwNP or other disease: Total number of SCS bursts per patient | From baseline up to 24 months.
Concomitant and prior medications for CRSwNP or other disease: Recovery of sense of smell after SCS | From baseline up to 24 months.
  Recovery of sense of smell after SCS will be described.
Concomitant and prior medications for CRSwNP or other disease:Time since the most recent SCS burst before initiation of Dupixent® | From baseline up to 24 months.
Concomitant and prior medications for CRSwNP or other disease: Number of prior or respiratory concomitant biotherapies per patient | From baseline up to 24 months.
  Number of prior, resp. concomitant biotherapies per patient
Concomitant and prior medications for CRSwNP or other diseases: Indication | From baseline up to 24 months.
  Indication (CRSwNP/Asthma/Atopic dermatitis/Prurigo nodularis/Eosinophilic esophagitis)
Concomitant and prior medications for CRSwNP or other diseases: Reason for stop | From baseline up to 24 months.
  Reason for stop will be describe.
Dupilumab (Dupixent®) modalities: Dosage | From baseline up to 24 months.
Dupilumab (Dupixent®) modalities: Injection modalities | From baseline up to 24 months.
  Injection modalities (Nurse/Caregiver/Self-injection)
Dupilumab (Dupixent®) modalities: Treatment duration | From baseline up to 24 months.
Dupilumab (Dupixent®) modalities: Compliance with treatment | From baseline up to 24 months.

SECONDARY OUTCOMES:
Change from baseline of Nasal polyps score (NPS) | From baseline up to 24 months
  The nasal polyps endoscopic score (NPS) assesses length and distribution of polyps, with a score from 0 to 4 for each nostril, maximum bilateral score of 8 points. Meaning lower (0=no polyp) and higher (4=large polyps).
Change from baseline of Nasal congestion score (NCS) | From baseline up to 24 months
  The Nasal congestion score (NCS) was assessed on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicating more severity.
Change from baseline of Smell test scores UPSIT | From baseline up to 24 months
  The UPSIT (UPSIT 40-odorant test) quantifies human olfactory function. Being the scores: ≤ 18 (anosmia) / [19-25] (severe hyposmia) / [26-30] (moderate hyposmia) / [31-34] (mild hyposmia) / [35-40] (normosmia)). A higher score indicating a better function.
Change from baseline of smell test score Visual Analog Scale (VAS) | From baseline up to 24 months
  Participants value their olfactory function by using the Visual Analogue Scale (VAS), the range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome), where higher score indicated worse thinkable troublesome.
Change from baseline of Quality of life questionnaire for patients with sino nasal symptoms (SNOT22) | From baseline up to 24 months
  SNOT-22 is a patient-reported outcome (PRO) questionnaire. Score ranges from 0 to 110 with higher score indicating greater rhinosinusitis related health burden.
Change from baseline of VAS for CRSwNP symptoms | From baseline up to 24 months
  The Visual Analog Scale for CRSwNP assesses symptoms, ranging from 0 to 10:
  * mild if VAS between 0 and 3
  * moderate if VAS between > 3 and 7
  * severe if VAS between > 7 and 10.
Change from baseline of Rhinorrhea score (anterior/posterior) | From baseline up to 24 months
  The rhinorrhea scores are scored from 0 ('No symptoms') to 3 ('Severe symptoms'). Where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicating more severity.
Change from baseline of number of SCS bursts/ surgery for CRSwNP | From baseline up to 24 months
  Rescue therapy: The number of SCS bursts/ surgery for CRSwNP will be reported.
Health care resource utilization (HCRU) for CRSwNP | From baseline up to 24 months.
  Health care resource utilization may include hospitalizations (including length of stay), outpatient visits, emergency room visits, specific transfusion visits.
Sense of smell impairment other than related to CRSwNP (Covid19) | From baseline up to 24 months.
  Collection of: Sense of smell impairment other than related to CRSwNP (Covid19) will be reported. If present, an Adverse Event (AE) will be recorded.
Number of Adverse Events (AE) / Serious Adverse Events (SAE) | From date of signed ICF or from date of Day 1 whichever comes first, up to 24 months
  The number of events and the percentage of patients who had at least one event will be described.
Site characteristics | At baseline (Day 1)
  Site characteristics (University/general Hospital/private clinic) will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number: 250.0001, Nantes, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org